CLINICAL TRIAL: NCT00519883
Title: Randomized Anastrozole Exercise Trial (The RAE Study)
Brief Title: Randomized Anastrozole Exercise Trial
Acronym: RAE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAE Study
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Musculoskeletal Symptoms
Keywords: Anastrozole; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Arm A: Standard Supportive Care (no supervised exercise)
  Interventions: Other: Supportive Care
- B (Experimental): Arm B: Exercise Intervention
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise
  Arms: B
Other: Supportive Care
  Arms: A

SUMMARY:
This is a randomized, phase III trial of a 12 week exercise program, followed by a 36 week voluntary, self-directed exercise program (total 48 weeks) compared to standard supportive care. The purpose of the trial is to determine whether the exercise program is better than standard supportive care to decrease the muscle and joint aches (musculoskeletal symptoms) that result from aromatase inhibitors.

Hypothesis An exercise program that includes stretching, strengthening and aerobic components may improve physical quality of life among women with musculoskeletal symptoms who are taking aromatase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Women who have been on an adjuvant AI for at least 6 weeks.
* The presence of some musculoskeletal symptoms.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1
* ER and or PgR positive early breast cancer, stages I, II or III
* Completion of any adjuvant chemotherapy (if given) and primary breast cancer surgery.
* Be willing to switch to Anastrozole if on another AI
* Signed written informed consent

Exclusion Criteria:

* Metastatic disease (no imaging or labs required in absence of clinical suspicion of metastases)
* Evidence or history of inflammatory arthropathy (for example, rheumatoid arthritis)
* Any medical condition (for example, significant heart disease) that would prevent a subject from completing an exercise program.
* Unable to take Aromatase Inhibitor (AI)
* Planned secondary reconstruction procedures during the 48 week study period
* Any medical, physical, geographic, emotional, or economic condition that in the judgement of the clinician/study doctor, would make an individual unable or unlikely to be able to exercise three times a week for 12 weeks.
* Unable to complete a study log book and questionnaires (unable to read and write English and no one at home who can adequately do so).
* The use of any exogeneous estrogen and/or progesterone except Estring and natural plant estrogens

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the mean SF36 physical component summary (PCS) score for subjects in each study Arm after 12 weeks.

SECONDARY OUTCOMES:
Difference in musculoskeletal symptoms as measured by VAS and NCIC-CTC toxicity criteria.
Global QOL: As measured by SF36 and VAS composite scores at each scheduled follow up visit (Baseline, weeks 4,8,12,24,36,48). See Appendix B for instruments.
Hot Flashes: A hot flash scale will be given to subjects to complete at each scheduled follow up visit (baseline, week 4,8,12,24,36,48). Severity and frequency of hot flashes will be compared between the exercise and control groups at each time point
Arm Circumferences: Arm circumferences will be measured for all subjects on both arms as described in Appendix D at each study follow up visit except weeks 4, 8, and 36.
Bone Mineral Density.
Body Mass Weight, in kilograms, will be recorded for all subjects at baseline and at weeks 4,8,12,24,36, and 48 week visits.

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Kennecke, MD, Principal Investigator — BC Cancer Agency Vancouver Centre; Caroline Lohrisch, MD, Principal Investigator — BC Cancer Agency - Vancouver Centre
Locations (2):
- Canada (2):
  - BC Cancer Agency Vancouver Centre, Vancouver, British Columbia
  - BC Cancer Agency Vancouver Island, Victoria, British Columbia